CLINICAL TRIAL: NCT07241182
Title: The Effects of Antrodia Cinnamomea Fruiting Body Extract on Quality of Life and Chemotherapy Side Effects in Patients With Lung Cancer Undergoing Platinum-Based Chemotherapy
Brief Title: Antrodia Cinnamomea Extract Effects on Lung Cancer Patients' Quality of Life During Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Collaborators: Balay Biotechnology Corporation (Unknown)
Responsible Party: Principal Investigator, Chen-Liang Tsai, Attending Physician, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A202505011
Record Dates: First submitted 2025-09-04; First posted 2025-11-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer (Diagnosis)
Keywords: Chemotherapy side effects; Lung cancer; Antrodia cinnamomea
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antrodia cinnamomea plus turmeric and probiotics (Experimental): Participants will receive capsules containing Antrodia cinnamomea extract, turmeric, and probiotics taken orally once daily for 3 months during platinum-based chemotherapy treatment.
  Interventions: Dietary Supplement: Antrodia cinnamomea supplement
- Turmeric and probiotics only (Active Comparator): Participants will receive capsules containing turmeric and probiotics (without Antrodia cinnamomea) taken orally once daily for 3 months during platinum-based chemotherapy treatment.
  Interventions: Dietary Supplement: Turmeric-Probiotic Group

INTERVENTIONS:
Dietary Supplement: Antrodia cinnamomea supplement — Intervention Description:
  Oral capsules containing Antrodia cinnamomea fruiting body extract combined with turmeric and probiotics, administered once daily for 3 months during platinum-based chemotherapy treatment. Each capsule contains standardized amounts of Antrodia cinnamomea extract, curcumin (from turmeric), and probiotic strains.
  Arms: Antrodia cinnamomea plus turmeric and probiotics
Dietary Supplement: Turmeric-Probiotic Group — Capsules containing turmeric and probiotics (without Antrodia cinnamomea), same dosing schedule and appearance as experimental group.
  Arms: Turmeric and probiotics only

SUMMARY:
This randomized trial will test whether Antrodia cinnamomea supplement improves quality of life in lung cancer patients receiving platinum-based chemotherapy.

Participants at Tri-Service General Hospital will be randomized to receive either Antrodia cinnamomea capsules or placebo for 3 months, with follow-up to 6 months (24 weeks). Primary outcomes include nausea/vomiting scores, sleep quality, quality of life, and cancer symptoms.

DETAILED DESCRIPTION:
This study will test whether a nutritional supplement, Antrodia cinnamomea can help improve quality of life in lung cancer patients receiving platinum-based chemotherapy.

Lung cancer patients often experience side effects from chemotherapy treatment, including nausea, vomiting, sleep problems, and other symptoms that affect their daily life. Antrodia cinnamomea is a medicinal mushroom supplement that may help reduce these side effects.

The study will include lung cancer patients who are receiving platinum-based chemotherapy at Tri-Service General Hospital. Participants will be randomly assigned to one of two groups: Participants will be randomly assigned to one of two groups: half will receive capsules containing turmeric, probiotics, and Antrodia cinnamomea, and half will receive capsules containing only turmeric and probiotics. Neither participants nor doctors will know which treatment each person is receiving.

All participants will take their assigned capsules daily for 3 months. Researchers will then continue to follow participants for an additional 3 months (up to 6 months total or 24 weeks) to monitor the lasting effects of the supplement. During this time, researchers will use questionnaires to measure nausea and vomiting, sleep quality, and cancer-related symptoms. The study will compare these measurements between the two groups to see if Antrodia cinnamomea supplement helps improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically and radio-graphically diagnosed lung cancer
* Age greater than 18 years
* Received platinum-based chemotherapy
* Life expectancy of six months or longer

Exclusion Criteria:

* Inability to comply with timely supplementation administration.
* Within 14 days prior to trial entry, laboratory data showing abnormal liver function, abnormal kidney function
* Within 30 days prior to trial entry, unexplained fever ≥38.5°C for 7 consecutive days or chronic diarrhea for 15 consecutive days.
* Currently receiving hormone therapy.
* Major cardiac disease or arrhythmia severe enough that the attending physician considers the patient unsuitable for trial participation.
* Major neuropathy.
* Patients with currently active acute infections.
* Patients with known allergies/allergic reactions to the investigational product or any components in their formulations.
* Patients currently taking supplements containing Antrodia camphorata extract.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Nausea and vomiting | Baseline, Week 3, Week 12, Week 18, and Week 24
  The Rhodes index of nausea, vomiting and retching (RINVR) will be used. While each item is scored from 0 to 4, the total possible score on the 8-item index is 32, with higher scores indicating greater severity.
Sleep quality | Baseline, Week 12, and Week 24
  Pittsburgh Sleep Quality Index (PSQI) will be used. Each component score of the PSQI ranges from 0 to 3, with the total possible score on the 7-component index being 21. The 0-3 scale assesses sleep dysfunction and disturbance, with higher scores indicating poorer sleep quality.
Symptom assessment | Baseline, Week 12, and Week 24
  The MD Anderson Symptom Inventory (MDASI) will be used. MDASI contains 19 items scored from 0 to 10, assessing symptom severity (13 items) and interference with daily activities (6 items). Higher scores indicate greater symptom burden.
Overall quality of life | Baseline, Week 12, and Week 24
  The EORTC QLQ-LC13 will be used. Each item on the 13-item EORTC QLQ-LC13 is scored from 1 to 4, assessing lung cancer-specific symptoms. Higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Skeletal muscle mass | Baseline, Week 3, Week 12, Week 18, and Week 24
  Skeletal muscle mass as measured by bioelectrical impedance analysis (BIA), reported in kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No